CLINICAL TRIAL: NCT02114996
Title: Phase 1 - Vocal Stimuli to Provoke Spontaneous Breathing
Brief Title: Can a Vocal Stimulus Provoke Spontaneous Breathing in an Ischemic Stroke Patient Dependent on Mechanical Ventilation?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Arnon Blum, Director of an Internal Medicine Department, The Baruch Padeh Medical Center, Poriya
Other Study IDs: B3072
Record Dates: First submitted 2014-04-13; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Patients Ventilated by Mechanical Ventilation With Ischemic Stroke
Keywords: mechanical ventilation; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Vocal stimulation may encourage spontaneous breathing in patients dependent on mechanical ventilation.

The study will include 30 patients on mechanical ventilation that will be intervened by the vocal stimulation and 30 patients on mechanical ventilation will serve as the control group.

DETAILED DESCRIPTION:
Vocal stimulation may encourage breathing in ventilated patients dependent on mechanical ventilation.

The study will include 30 patients on mechanical ventilation that will be intervened by the vocal stimulation and 30 patients on mechanical ventilation that will be our control group.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke men and women older than 18 years old and younger than 80 years old

Exclusion Criteria:

* coma from other reasons other than ischemic stroke hemmorhagic stroke active malignancy renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients on mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
spontaneous breathing | 3 days
  we anticipate a better response and recurring spontaneous breathing in the treatment group.